CLINICAL TRIAL: NCT01493674
Title: Folic Acid Supplementation for Improving Homocysteine Levels, Cognitive and Depressive Status in Eating Disorders
Brief Title: Folic Acid Supplementation in Eating Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Principal Investigator, Ignacio Galicia, Head of Research and Clinical Trial Department, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HULP 2448; 2007-004353-28 (EudraCT Number)
Record Dates: First submitted 2011-12-13; First posted 2011-12-16 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Eating Disorders
Keywords: folate; homocysteine; cognitive function; eating disorders; depression.
MeSH Terms: conditions — Feeding and Eating Disorders; Depression | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo tablets (No Intervention): two identical tablets, but composed of crystalline cellulose, lactose and colouring
- a suplemented group (Experimental): two 5-mg tablets of folic acid
  Interventions: Dietary Supplement: folic acid

INTERVENTIONS:
Dietary Supplement: folic acid — two 5-mg tablets of folic acid
  Other Names: folic acid (ACFOL®)
  Arms: a suplemented group

SUMMARY:
The aim of this study was to determine the effect of folic acid supplementation on homocysteine levels in a group of patients with eating disorders (ED) with low folate intake. The secondary aims were to evaluate the evolution on cognitive and depressive status after the intervention.

DETAILED DESCRIPTION:
Some authors have identified the presence of increased levels of homocysteine in patients with eating disorders and attempts have been made to find some association between this and the high rates of depression and cognitive function impairment recorded in these patients. It is still not known what causes this increase in homocysteine levels, whether the levels return to normal after the nutritional state is normalised and what strategies must be employed to carry out this normalisation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females diagnosed with eating disorders (DSM-IV criteria of the American Psychiatric Association, 2000)
* Age > 18 years
* Low folate intake based on the recommended daily intake in terms of age (Institute of Medicine, 1998)

Exclusion Criteria:

* Patients with contraindications for folic acid supplementation due to hypersensitivity to folic acid or anaemia due to lack of B12
* Patients who routinely used drugs that interfere with folic acid absorption (analgesics, anticonvulsants, hydantoin, carbamazepine, antacids, antibiotics, cholestyramine, methotrexate, pyrimethamine, triamterene, trimethoprim and sulphonamides)
* Patients with vitamin and mineral supplements intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Blood variables monitored | after 6 month of intervention
  serum folate, red blood cell folate, vitamin B12, plasma homocysteine

SECONDARY OUTCOMES:
Evolution on cognitive and depressive status | after 6 month of intervention
  Beck Depression Inventory Test Stroop colour-word interference test Trail Making Test
Anthropometric parameters | after 6 month of intervention
  weight, body composition, food frequency questionnaire
Dietary parameters | after 6 months of intervention
  Energy, macronutrients and micronutrients intake.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, MD, Principal Investigator — Nutrition Department. La Paz University Hospital. La Paz Health Research Institute.
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain